CLINICAL TRIAL: NCT02780466
Title: Observational Study on Intubation in Septic Shock
Acronym: INTUBATIC
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Principal Investigator, DENISE JOLIVOT, Coordinator for medical research, University Hospital, Angers
Other Study IDs: 2015-96
Record Dates: First submitted 2016-05-19; First posted 2016-05-23 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Septic Shock
Keywords: Septic shock; Endotracheal intubation; Outcome
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients with septic shock

SUMMARY:
Septic shock is common in intensive care and its mortality remains high. While new treatments have not improved survival, optimization of known and widely used techniques has allowed reduction in mortality. Thus improving care given to patients starts with making better use of existing resuscitation techniques. Among these practices, mechanical ventilation is widespread in the management of patients with septic shock. In large studies published in recent years in Europe and North America, 40 to 85% of patients receive invasive mechanical ventilation. It therefore appears that a significant proportion of patients are never intubated during treatment and management of their septic shock. There is no specific recommendation from critical care societies concerning mechanical ventilation in the treatment of septic shock. Apart from indisputable situations such as impaired consciousness or acute respiratoire distress, the decision whether to ventilate mechanically or not is left to the discretion of the physician.

The aim of this study is to analyze intubation practice in septic shock patients and its impact on 28-day survival.

This multicentric and observational study will be conducted in 30 French ICUs.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years old
* Admitted in the ICU for septic shock
* Introduction of vasopressors ( norepinephrine or adrenaline ) in the ICU or within 24 hours of ICU admission
* Suspected or proven infection

Exclusion Criteria:

* Intubation before the introduction of vasopressors
* Decision of withdrawing or withholding care at admission
* Pregnant woman
* Patient not affiliated to the social security insurance
* Refusal of participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in the study are adults patients admitted to intensive care unit in France (about 30 centers) for shock, supposed or confirmed of septic origin.
Sampling Method: Non-Probability Sample
Enrollment: 859 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
death | 28 days after ICU admission

SECONDARY OUTCOMES:
duration of organ support | 28 days
  mechanical ventilation, vasopressors, renal replacement therapy
impact of intubation delay on outcome | 28 days

REFERENCES:
- [Derived] Mellado-Artigas R, Ferrando C, Martino F, Delbove A, Ferreyro BL, Darreau C, Jacquier S, Brochard L, Lerolle N. Early intubation and patient-centered outcomes in septic shock: a secondary analysis of a prospective multicenter study. Crit Care. 2022 Jun 7;26(1):163. doi: 10.1186/s13054-022-04029-6. PMID 35672860
- [Derived] Darreau C, Martino F, Saint-Martin M, Jacquier S, Hamel JF, Nay MA, Terzi N, Ledoux G, Roche-Campo F, Camous L, Pene F, Balzer T, Bagate F, Lorber J, Bouju P, Marois C, Robert R, Gaudry S, Commereuc M, Debarre M, Chudeau N, Labroca P, Merouani K, Egreteau PY, Peigne V, Bornstain C, Lebas E, Benezit F, Vally S, Lasocki S, Robert A, Delbove A, Lerolle N. Use, timing and factors associated with tracheal intubation in septic shock: a prospective multicentric observational study. Ann Intensive Care. 2020 May 24;10(1):62. doi: 10.1186/s13613-020-00668-6. PMID 32449053